CLINICAL TRIAL: NCT06312709
Title: teleABLE: Adapting a Behavioral Activation-Based Intervention to Reduce Post-Stroke Sedentary Behavior Using Telehealth (Pilot Randomized Controlled Trial)
Brief Title: teleABLE to Reduce Post-Stroke Sedentary Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00021288; K23HL159240 (NIH)
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Stroke
Keywords: sedentary behavior; physical activity; behavioral activation; activity engagement; occupational therapy; rehabilitation
MeSH Terms: conditions — Stroke; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- teleABLE (Experimental): Participants meet with a study therapist 2x/week for 6 weeks (12 sessions) to complete behavioral activation focused on adding personally meaningful non-sedentary activities during times when they typically spend sitting. All sessions are delivered remotely using Zoom videoconferencing.
  Interventions: Behavioral: teleABLE (telehealth-delivered Activating Behavior for Lasting Engagement)
- Health Education (Active Comparator): Participants meet with a study therapist 1x/week for 6 weeks (6 sessions) to review fact sheets focused on healthy lifestyles after stroke. All sessions are delivered remotely using Zoom videoconferencing.
  Interventions: Other: Health Education

INTERVENTIONS:
Behavioral: teleABLE (telehealth-delivered Activating Behavior for Lasting Engagement) — teleABLE uses behavioral activation to build personally meaningful non-sedentary throughout the day. This is accomplished using a global strategy, the ICAN Planning Process, which guides participants through activity scheduling, activity monitoring, self-assessment, and collaborative problem solving.
  Arms: teleABLE
Other: Health Education — Health Education provides information about stroke using factsheets from the American Heart Association and reflection questions that support participants in applying the information.
  Arms: Health Education

SUMMARY:
The goal of this clinical trial to test whether a remotely delivered behavioral activation-based intervention called "teleABLE" works better than a health education intervention for (1) reducing sitting time and (2) improving health-related quality among adults who were diagnosed with stroke within the past 12 months.

Participants in this study will:

* Complete questionnaires at Weeks 1, 8, and 24
* Wear an activPAL monitor at Weeks 1, 8, and 24
* Participate in the teleABLE intervention (12 sessions) or the health education intervention (6 sessions)
* Complete an interview at Week 24

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Diagnosis: Stroke diagnosis ≤12 months prior to study enrollment
* ≥6 hours of sedentary behavior on a typical weekday (Sedentary Behavior Questionnaire)
* Able to walk 150 feet or more without physical assistance from another person, with or without assistive device (assessed by Functional Independence Measure, mobility score ≥5)
* Able to access an electronic device (smartphone, tablet, or computer) that is compatible with a videoconferencing application
* Able to identify a support person with whom they have a face-to-face interaction at least one time per week.
* Able and willing to participate fully in the study and provide informed consent

Exclusion Criteria:

* Currently receiving care in an inpatient rehabilitation, transitional care unit, or skilled nursing facility
* Severe cognitive or communication impairments (inability to respond accurately to complete study telephone screening or complete informed consent)
* Comorbid neurodegenerative disorder (e.g. Parkinson's disease, multiple sclerosis, amyotrophic lateral sclerosis, myasthenia gravis, dementia, Alzheimer's disease, Huntington's disease, glioblastoma)
* Comorbid cancer, currently undergoing chemotherapy or radiation treatment
* Comorbid major depressive disorder (Patient Health Questionnaire-2, score ≥2)
* Received inpatient treatment or hospitalized for psychiatric condition and/or alcohol or substance abuse within the past 12 months
* Diagnosis of a terminal illness and/or currently receiving hospice care
* Currently pregnant or expecting to become pregnant in the next 6 months
* History of skin sensitivity that precludes the use of medical tape necessary for adherence to activity monitor measure
* Inability to speak, read, or understand English
* Concurrent participation in any other rehabilitation intervention research study (including cognitive and/or physical rehabilitation studies)
* Investigator discretion for safety or adherence reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in change scores on health-related quality of life | Week 0 to Week 8
  European Quality of Life 5-Dimension 5-Level (EuroQOL-5D-5L) change score. The possible range on this tool is -1 (worst) to 1 (best).
Between-group difference in change in sedentary behavior | Week 0 to Week 8
  Change in mean minutes per day spent in prolonged sedentary time (accumulated in bouts of 30 minutes or more) measured using the activPAL micro4 (7-day wear protocol)

SECONDARY OUTCOMES:
Between-group difference in change in sedentary behavior | Week 0 to Week 24
  Change in mean minutes per day spent in prolonged sedentary time (accumulated in bouts of 30 minutes or more) measured using the activPAL micro4 (7-day wear protocol)
Between-group difference in change scores on health-related quality of life | Week 0 to Week 24
  European Quality of Life 5-Dimension 5-Level (EuroQOL-5D-5L) change score. The possible range on this tool is -1 (worst) to 1 (best).

OTHER OUTCOMES:
Between-group difference in change in step count | Week 0 to Week 8
  Mean daily step count measured using the activPAL micro4 (7-day wear protocol)
Between-group difference in change in step count | Week 0 to Week 24
  Mean daily step count measured using the activPAL micro4 (7-day wear protocol)
Between-group difference in change in total activity retention | Week 0 to Week 8
  Change in the proportion of total activities retained measured using the Activity Card Sort (ACS3)
Between-group difference in change in total activity retention | Week 0 to Week 24
  Change in the proportion of total activities retained measured using the Activity Card Sort (ACS3)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Kringle, PhD, OTR/L, Principal Investigator — University of Minnesota
Locations (1):
- School of Kinesiology, University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No